CLINICAL TRIAL: NCT00669383
Title: Rescue Antenatal Steroids and Lung Volumes in Preterm Infants
Brief Title: Rescue Antenatal Steroids and Pulmonary Function Tests in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Cynthia McEvoy, Associate Professor of Pediatrics, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OHSU eRIB#1845
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Compliance; Functional Residual Capacity; Pulmonary Function Testing
Keywords: premature delivery; respiratory distress syndrome
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Betamethasone (Celestone) 12 mg intramuscular q 24 hours x 2 doses
  Interventions: Drug: betamethasone
- B (Placebo Comparator): Placebo dose intramuscular q 24 hours x 2 doses
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: betamethasone — 12 mg IM q 24 hours x 2 doses
  Other Names: Celestone
  Arms: A
Drug: placebo — Placebo IM q 24 hours x 2 doses
  Arms: B

SUMMARY:
One course of steroids given to a mother before a premature delivery helps the lungs of the premature infant and decreases breathing problems. One course of antenatal steroids is the standard of care for threatened premature deliveries. It is unclear as to how long the benefit of one course of steroids last. The most benefit to the baby's lungs seem to occur if the steroids are given at least 24 hours before but within 7 days of a premature delivery. It is difficult to predict the timing of a preterm delivery so deliveries often do not occur within this time period. We hypothesize that the benefits of the steroids to the lungs wear off if the steroids are given more than 14 days before a preterm delivery, and that in these circumstances an extra course of steroids will help the premature baby's lungs and the premature baby will have less breathing problems as shown by lung function testing.

DETAILED DESCRIPTION:
The primary purpose of this randomized, blinded placebo controlled trial is to quantify and compare measurements of pulmonary function (including respiratory compliance and lung volumes/functional residual capacity) of hospitalized preterm infants whose mothers received an initial course of antenatal corticosteroids, remained undelivered after 14 days and at < 34 weeks of gestation, and were then randomized to either a rescue course of antenatal corticosteroids or to a rescue course of placebo. In addition, follow-up pulmonary function tests, clinical outcomes, growth parameters, and the neurodevelopmental outcome of these infants will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 14 days after first course of antenatal steroids;
* Less than 34 weeks of gestation;
* Identified by primary physician as continued risk for preterm delivery;
* Informed consent

Exclusion Criteria:

* Major congenital anomalies
* Multiple gestation of triplets or greater
* Mother with insulin dependent diabetes

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2001-06; Primary Completion 2007-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia McEvoy, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] McEvoy C, Schilling D, Peters D, Tillotson C, Spitale P, Wallen L, Segel S, Bowling S, Gravett M, Durand M. Respiratory compliance in preterm infants after a single rescue course of antenatal steroids: a randomized controlled trial. Am J Obstet Gynecol. 2010 Jun;202(6):544.e1-9. doi: 10.1016/j.ajog.2010.01.038. Epub 2010 Mar 15. PMID 20227053
- [Result] McEvoy C, Schilling D, Spitale P, O'Malley J, Bowling S, Durand M. Pulmonary function and outcomes in infants randomized to a rescue course of antenatal steroids. Pediatr Pulmonol. 2017 Sep;52(9):1171-1178. doi: 10.1002/ppul.23711. Epub 2017 Apr 24. PMID 28436580
- [Result] Jordan BK, Schilling D, McEvoy CT. The window of improved neonatal respiratory compliance after rescue antenatal steroids. J Perinatol. 2018 Jul;38(7):828-833. doi: 10.1038/s41372-018-0124-9. Epub 2018 May 24. PMID 29795314
- [Result] Jordan BK, Schilling D, McEvoy CT. Pulmonary Function at Hospital Discharge in Preterm Infants Randomized to a Single Rescue Course of Antenatal Steroids. J Pediatr. 2017 Feb;181:62-66.e1. doi: 10.1016/j.jpeds.2016.10.022. Epub 2016 Nov 7. PMID 27832835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized trial was conducted at Oregon Health and Science University in Portland, OR and at Sacred Heart Hospital in Pensacola, FL. Subjects were recruited from June 2001 to May 2007.
Pre-assignment Details: Women who showed no further signs of preterm delivery after consent were not randomized.
Groups:
- A (Betamethasone): Betamethasone (Celestone) 12 mg IM q 24 hours x 2 doses
- B (Placebo): Placebo dose IM q 24 hours x 2 doses
Period: Overall Study
Arm/Group | A (Betamethasone) | B (Placebo)
Started | 44 | 41
Completed | 44 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A (Betamethasone): Betamethasone (Celestone) 12 mg IM q 24 hours x 2 doses
  betamethasone: 12 mg IM q 24 hours x 2 doses
- B (Placebo): Placebo dose IM q 24 hours x 2 doses
  placebo: Placebo IM q 24 hours x 2 doses
- Total: Total of all reporting groups
Arm/Group | A (Betamethasone) | B (Placebo) | Total
Number analyzed (Participants) | 44 | 41 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 41 | 85
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 26.9 (7.5) | 28.6 (6.4) | 27.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 41 | 85

OUTCOME MEASURES:

1. Primary Outcome: Measurements of Functional Residual Capacity in Preterm Infants.
Time Frame: Within first 72 hours after birth
Population: Number of participants listed here is greater than the number listed in Participant flow as twin deliveries were not excluded.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | A (Betamethasone) | B (Placebo)
Number analyzed (Participants) | 49 | 49
mL/kg | 24.8 (8.8) | 22.0 (7.9)

2. Primary Outcome: Measurements of Respiratory Compliance (Crs) in Preterm Infants.
Time Frame: Within first 72 hours after birth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/cm H2O/kg
Arm/Group | A (Betamethasone) | B (Placebo)
Number analyzed (Participants) | 49 | 49
mL/cm H2O/kg | 1.21 (0.53) | 1.01 (0.51)

3. Secondary Outcome: FiO2
Time Frame: During initial hospital stay and planned follow-up
Population: Number of participants is greater here as it includes all offspring, including twins.
Measure: Count of Participants; unit: Participants
Arm/Group | A (Betamethasone) | B (Placebo)
Number analyzed (Participants) | 56 | 56
Participants
  FiO2 greater or equal to 0.30 | 7 | 16
  FiO2 greater or equal to 0.40 | 5 | 13

ADVERSE EVENTS:
Description: Number of participants listed here is greater than the number listed in participant flow as this section includes offspring and twins were included.
Arm/Group | A (Betamethasone) | B (Placebo)
All-Cause Mortality (participants affected / at risk) | 1/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No